CLINICAL TRIAL: NCT00194285
Title: FDG-PET Imaging in Painful Joint Prosthesis (Protocol Amendment, Version 11, Dated 9/2005)
Brief Title: FDG-PET Imaging in Painful Joint Prosthesis
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01AR048241-03 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Painful Joint Prostheses
Keywords: Prosthesis; [18 F] Fluorodeoxyglucose; Positron Emission Tomography Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: FDG-PET Imaging

SUMMARY:
The main objective of the proposed research study is to determine the efficacy of [18-F] Fluorodeoxyglucose (FDG) positron emission tomography (PET) in differentiating infections from other complications such as loosening in patients with painful joint prosthesis. We intend to validate and establish the necessary criteria for making such a diagnosis and determine the accuracy of the technique through comparison with other existing modalities such as white blood imaging and patient outcome. We expect that at the completion of the proposed research, the role of this novel and powerful imaging modality will be clearly defined in the management of patients with this challenging and serious complication.

DETAILED DESCRIPTION:
The purposes of this study are: 1. To determine the normal pattern of FDG uptake demonstrated by pet up to two years following total joint replacement surgery 2. To establish the optimal diagnostic criteria for differentiating septic from aseptic painful joint prosthesis by FDG-PET imaging and determine its accuracy 3. To compare the accuracy of FDG-PET imaging to conventional techniques for the differentiation of septic from aseptic painful joint prostheses.

We intend to enroll 100 patients per year for 5 years. These patients will be selected from more than 300 cases that undergo joint revisions at the collaborating institutions. After each patient undergoes an appropriate evaluation including history, physical examination, radiographic and laboratory evaluation, he/she will be assigned into one of the groups listed below based on the degree of suspicion of an infectious process. Every effort will be made to have approximately one-third of the patients recruited from each of the following groups.

Study Plan Study I: FDG-PET imaging in the painful partial or total joint prosthesis We intend to enroll 100 patients per year for 5 years. These patients will be selected from more than 300 cases that undergo joint revisions at the collaborating institutions. After each patient undergoes an appropriate evaluation including history, physical examination, radiographic and laboratory evaluation, he/she will be assigned into one of the groups listed below based on the degree of suspicion of an infectious process. Every effort will be made to have approximately one-third of the patients recruited from each of the following groups.

Group 1: Low pre-scan suspicion of infection. The incidence of infection based on past experience is <10% in this population.

Group 2: High pre-scan suspicion of infection. The incidence of infection in this group is quite high based on past experience.

Group 3: Intermediate pre-scan suspicion of infection. Criteria: Any patient who does not fit into either group 1 or 2 will be considered for this category. The incidence of infection in this group based on past experience is intermediate.

Considering the large number of patients who undergo joint revision (more than 300 annually) in the participating institutions combined, we expect no difficulties in recruiting adequate numbers in all 3 categories.

Each patient will undergo only one preoperative diagnostic FDG-PET scan. After the PET scan is completed, a diagnosis and detailed description of the observations made will be communicated to the attending surgeon before the operation. We believe this information will enable investigators to establish the correct diagnosis during surgical intervention.

Study II: FDG-PET imaging following uncomplicated partial or total joint arthroplasty To accomplish this goal, we will enroll 10 patients per year for the first 3 years. FDG-PET scans will be performed at approximately 12 months, 18 months and/or 2 years following surgery. All scans will occur within 2 months of the 12-, 18-, and/or 24-month anniversary of that patient's most recent joint replacement surgery. It is unknown how long FDG uptake persists in an uncomplicated partial or total joint arthroplasty. The expected pattern of FDG uptake following arthroplasty will provide a basis for the correct diagnosis of periprosthetic infection and loosening during the life of the implant.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected for entry into this study will be men or women of any ethnic background who are scheduled to undergo clinical and diagnostic evaluation by a member of the Department of Orthopedic Surgery at the Hospital of the University of Pennsylvania Health System or by the collaborating physicians at the Rothman Institute or the VA Philadelphia Medical Center.

Study I: FDG-PET imaging in painful partial or total joint prostheses Each patient who is a candidate will be evaluated by one of the collaborators mentioned above for a painful partial or total joint prosthesis. The patient will undergo an appropriate routine evaluation including history, physical examination, radiographic, scintigraphic, and necessary laboratory evaluation. An initial diagnosis must be made for each patient. The diagnosis of loosening will be established based on clinical examination and/or radiographic evaluation demonstrating clear evidence of this complication. Other etiologies for the joint pain, except for infection and aseptic loosening, need to be excluded. Surgical intervention (prosthesis revision) may or may not be planned for the patient who is a candidate for this study.

Study II: FDG-PET imaging following uncomplicated partial or total joint arthroplasty All patients fulfilling the criteria below will be considered potential candidates for this study. Each patient must have a diagnosis of degenerative joint disease caused by osteoarthritis (no previous hip surgery) and have undergone primary partial or total joint arthroplasty by a member of the Department of Orthopedic Surgery at the Hospital of the University of Pennsylvania or referring hospitals. Other causes of degenerative joint disease will be excluded by physical, radiographic and laboratory evaluation as clinically indicated. Osteoarthritis is the most common cause of degenerative joint disease, and in order to avoid any confounding factors in experimental results that may be caused by other types of disorders, only this group of patients will be studied. A patient will be eliminated from this group at anytime if the post-operative course is complicated by any process that is thought to influence the outcome. Variations from an uncomplicated postoperative course will be determined by the operating surgeon and include clinical signs or other evidence to suggest infection, early loosening, or any other process directly involving the prosthesis.

Exclusion Criteria:

* Patients with other etiologies for pain, other than for infection and aseptic loosening, will be excluded from enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Five hundred patients selected for entry into this study will be men or women of any ethnic background who are scheduled to undergo clinical and diagnostic evaluation for joint prosthesis revision by members of the Department of Orthopedic Surgery at the University of Pennsylvania Health System (Hospital of University of Pennsylvania and Pennsylvania Hospital) or by the collaborating physicians at the Rothman Institute at Thomas Jefferson University Hospital or the VA Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2001-03; Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
SUV measurement from PET scan | Assessed after FDG scan
  Standardized Uptake Value

CONTACTS AND LOCATIONS:
Overall Officials: Abass Alavi, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States